CLINICAL TRIAL: NCT00409656
Title: Prospective, Randomized Trial of Basiliximab (Simulect) in the Prophylaxis of High-Risk Keratoplasty Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FR-2003-12-2005-12
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2006-12-13 (Estimated); Status verified 2006-12

CONDITIONS: Corneal Transplantation
MeSH Terms: interventions — Basiliximab

INTERVENTIONS:
Drug: Basiliximab

SUMMARY:
Most high risk keratoplasties are currently performed under systemic immunosuppression. Immunosuppressants are currently either Cyclosporine A or mycophenolate mofetile, administered for around 6 months. Due to potentially severe adverse effects, new immunosuppressive exerting less side effects would be desirable. Basiliximab is a monoclonal, chimeric antibody, targeted specifically against the Interleukin-2-Rezeptor from activated T-cells. This agent is known to specifically inhibit T-cell proliferation upon intravenous application only twice following transplantation. Basiliximab has already been demonstrated effective in kidney transplantation.

This investigation is a prospective, randomized clinical trial on orthotopic, high-risk penetrating keratoplasty. Basiliximab is evaluated against systemic Cyclosporine A. Primary endpoint is graft rejection. Secondary endpoint is clear graft survival.

ELIGIBILITY:
Inclusion Criteria:

* high risk keratoplasty

Exclusion Criteria:

* normal risk keratoplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-12; Study Completion 2005-12

PRIMARY OUTCOMES:
Graft rejection

SECONDARY OUTCOMES:
Clear graft survival

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Reinhard, MD, Prof., Study Director — University Eye Hospital, Freiburg

REFERENCES:
- [Derived] Abudou M, Wu T, Evans JR, Chen X. Immunosuppressants for the prophylaxis of corneal graft rejection after penetrating keratoplasty. Cochrane Database Syst Rev. 2015 Aug 27;2015(8):CD007603. doi: 10.1002/14651858.CD007603.pub2. PMID 26313245